CLINICAL TRIAL: NCT00337298
Title: Lack of Effect of Antihypertensive Treatment With Amlodipine and Lisinopril on Retinal Autoregulation in Patients With Type 1 Diabetes and Mild Diabetic Retinopathy. A Prospective Randomized Clinical Trial.
Brief Title: The Effect of Amlodipine and Lisinopril on Retinal Autoregulation in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Velux Fonden (Other)
Responsible Party: Toke Bek/Professor, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: Jmehl01
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Type 1 Diabetes; Diabetic Retinopathy; Eye Diseases; Diabetes Complications
Keywords: Diabetes; Retinopathy; Blood Pressure; Amlodipine; Lisinopril
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy; Eye Diseases; Diabetes Complications; Diabetes Mellitus; Retinal Diseases | interventions — Amlodipine; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Crossover design. Arm is same all the way
  Interventions: Drug: Amlodipine; Drug: Lisinopril

INTERVENTIONS:
Drug: Amlodipine — 1 (5mg) tablet daily, given 14 days totally before measure of outcome.
Drug: Lisinopril — Lisinopril 10 mg given daily for 14 days and then outcome was measured.

SUMMARY:
The purpose of this study is to compare the effect of two antihypertensive drugs on retinal vessel diameter in young type 1 diabetics. The retinal vessel analyzer (RVA) was used to investigate how the drugs affected vessel diameter, when the subjects were exposed to an increase in blood pressure, induced by isometric muscle contraction and when they were stimulated by flickering light.

DETAILED DESCRIPTION:
Diabetes is a leading cause of blindness in the western part of the world. Diabetic patients develop diabetic retinopathy which can progress to blindness. Diabetic retinopathy is associated with an increase of blood flow in the retinal vessels, ischaemia in the periphery and macular oedema. It has been shown in previous trials, that the pressure and metabolic autoregulation is disturbed in patients with diabetes, and it is believed to contribute to the development of diabetic retinopathy.

In healthy subjects the retinal arterioles will contract during an increase in blood pressure, but trials have shown that this response is impaired in diabetics. When the retina is exposed to flickering lights, the metabolism increase and the arterioles in healthy subjects dilates. In diabetics this dilation is impaired. In this trial we want to investigate if an ACE-inhibitor (lisinopril) or calcium channel blocker (amlodipine) influence this response in subjects exposed to increased blood pressure vs increased retinal metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* 18-35 years of age
* Simplex retinopathy at last screening (Less than 10 retinal haemorrhages at the nearest ordinary screening examination)
* normotensive (BP not above 160 mmHg systolic or 100 mmHg diastolic)

Exclusion Criteria:

* Pregnancy
* Systolic Bloodpressure above 160 mmHg
* Diastolic bloodpressure above 100 mmHg
* Retinopathy grade higher than simplex retinopathy
* Prior retinal laser photocoagulation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Vessel diameter changes in arbitrary units as measured with the Retinal Vessel Analyzer | 120,240,360,480,600,720 and at 840secs

SECONDARY OUTCOMES:
Blood pressure (mmHG) | 120,240,360,600,720,840 secs
24 hour ambulatory blood pressure (mmHg) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Toke Bek, MD, PhD, Principal Investigator — Aarhus university hospital, Dep. of ophthalmology; Per L Poulsen, MD, PhD, Principal Investigator — Aarhus University hospital, Dep. of endocrinology (M)
Locations (1):
- Aarhus university hospital, Aarhus, Denmark